CLINICAL TRIAL: NCT00900380
Title: Comparison of P-gp Efflux and Accumulation Assay Results With ECOG 3999 Leukemia Samples
Brief Title: Studying Tissue Samples to Learn More About Drug Resistance in Patients With Acute Myeloid Leukemia
Status: Completed | Type: Observational
Sponsor: ECOG-ACRIN Cancer Research Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: Eastern Cooperative Oncology Group (Network)
Other Study IDs: CDR0000478869; ECOG-E3999T1
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2017-05-19 (Actual); Status verified 2017-05

CONDITIONS: Leukemia
Keywords: adult acute monocytic leukemia (M5b); adult acute megakaryoblastic leukemia (M7); adult acute myeloblastic leukemia with maturation (M2); adult acute myeloblastic leukemia without maturation (M1); adult acute myelomonocytic leukemia (M4); adult acute monoblastic leukemia (M5a); secondary acute myeloid leukemia; untreated adult acute myeloid leukemia; adult acute minimally differentiated myeloid leukemia (M0); adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); adult erythroleukemia (M6a); adult pure erythroid leukemia (M6b)
MeSH Terms: conditions — Leukemia; Leukemia, Monocytic, Acute; Leukemia, Megakaryoblastic, Acute; Leukemia, Myeloid, Acute; Leukemia, Myelomonocytic, Acute; Congenital Abnormalities; Leukemia, Erythroblastic, Acute | interventions — Flow Cytometry

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective

INTERVENTIONS:
Other: flow cytometry
Other: immunological diagnostic method
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying samples of tissue from patients with cancer in the laboratory may help doctors learn more about cancer and the development of drug resistance in patients.

PURPOSE: This laboratory study is examining tissue samples from patients with acute myeloid leukemia to learn more about drug resistance in these patients.

DETAILED DESCRIPTION:
OBJECTIVES:

* Ascertain whether assessments of P-glycoprotein (P-gp) status using the accumulation assay find greater than 10% positive specimens among 30 specimens (collected from patients with acute myeloid leukemia enrolled on clinical trial ECOG-E3999) found to be negative using only the efflux assay.

OUTLINE: This is a multicenter study.

Cryopreserved bone marrow specimens are examined for P-glycoprotein (P-gp) by the accumulation assay and the efflux assay using DiOC_2 dye. Flow cytometry is used for measuring activity in both assays.

PROJECTED ACCRUAL: A total of 40 specimens will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Cryopreserved bone marrow specimens collected from patients with acute myeloid leukemia enrolled on clinical trial ECOG-E3999 meeting the following criteria:

  * Appreciable levels of either CD34+ OR CD117+ blasts
  * Appreciable staining with anti-P-gp antibodies
* 30 specimens must exhibit low to moderate dye loading for the Rh123 efflux assay
* 10 specimens must exhibit positive Rh123 efflux activities

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Samples submitted for research from patients participating in E3999
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2006-03-28 (Actual); Primary Completion 2013-12-30 (Actual); Study Completion 2013-12-30 (Actual)

PRIMARY OUTCOMES:
Percentage of specimens collected from patients that are found to be P-glycoprotein (P-gp)-positive by accumulation assay that were found to be negative using efflux assay | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Paietta, PhD, Study Chair — Our Lady of Mercy Medical Center